CLINICAL TRIAL: NCT01227759
Title: A Phase IIa, Single-center, Randomized, Observer-blind Trial With Intraindividual Comparison of Treated Versus Untreated to Assess the Wound Healing Efficacy of Topical Tyrosur® Gel
Brief Title: Tyrosur® Gel-Investigation on Wound Healing Efficacy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Engelhard Arzneimittel GmbH & Co.KG (Industry)
Responsible Party: W. Wigger-Alberti, M.D., bioskin GmbH
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EA-10-1-042
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Wounds; Wound Healing
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Verum (Experimental)
  Interventions: Drug: Drug containing the active ingredient
- Untreated (No Intervention)
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug containing the active ingredient — The topical application is performed once daily during a 12-day treatment.
  Other Names: Tyrosur® Gel
  Arms: Verum
Drug: Placebo — Placebo containing no active ingredient
  Other Names: Vehicle to Tyrosur® Gel
  Arms: Vehicle

SUMMARY:
This IIa study with intraindividual comparison of treated versus untreated to assess the wound healing efficacy of Tyrosur® Gel after experimental impairment of the skin using an abrasive wound healing model.

DETAILED DESCRIPTION:
This is a single-center, randomized, observer-blind phase IIa study with intraindividual comparison of treated versus untreated to assess the wound healing efficacy of Tyrosur® Gel after experimental impairment of the skin using an abrasive wound healing model.

In the investigation two small, superficial, abrasive wounds will be induced on the right forearm and one on the left forearm of each subject using a sterile surgical hand brush. These wounds will then be treated with the investigational products. The wound healing will be clinically assessed and photographs will be taken for documentation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older with healthy skin in the test area
* The physical examination must be without disease findings unless the investigator considers an abnormality to be irrelevant for the outcome of the clinical trial;
* Written informed consent obtained.

Exclusion Criteria:

* acne, suntan, eczema, hyperpigmentation or tattoos in the test fields;
* dark-skinned persons whose skin color prevents ready assessment of skin reactions;
* subjects with diabetes, psoriasis or lichen ruber planus;
* history of wound-healing complications, or keloid and hypertrophic scarring;
* evidence of drug or alcohol abuse;
* pregnancy or nursing;
* symptoms of a clinically significant illness that may influence the outcome of the trial in the four weeks before and during the trial;
* known allergic reactions to components of the investigational product/s;
* treatment with systemic or locally acting medications which might counter or influence the trial aim within two weeks before the baseline visit (e.g. antihistamines or glucocorticosteroids);
* contraindications according to summary of product characteristics;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of the wound healing efficacy of verum compared to untreated using a score for wound healing rates | 12 days

SECONDARY OUTCOMES:
Clinical assessment of the wound healing efficacy of the vehicle compared to untreated using a score for wound healing rates; Photo documentation of the wound healing efficacy | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Walter Wigger-Alberti, MD, Principal Investigator — Managing director bioskin, Hamburg Germany